CLINICAL TRIAL: NCT07245524
Title: PeriOPerative Spine Surgery COntrol Pain (POPSSCOP) Study: Intrathecal Morphine vs Erector Spinae Plane Block for Postoperative Pain Management in Spinal Fusion. Single-center Prospective Observational Study
Brief Title: PeriOPerative Spine Surgery COntrol Pain (POPSSCOP) Study: Intrathecal Morphine vs Erector Spinae Plane Block for Postoperative Pain Management in Spinal Fusion
Acronym: POPSSCOP
Status: Completed | Type: Observational
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Sponsor
Other Study IDs: 210/2024
Record Dates: First submitted 2025-09-30; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Spine Fusion; Locoregional Anaesthesia; Intrathecal Anesthesia; Erector Spina Plan Block; Multimodal General Anesthesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IM: Intrathecal Morphine: Patients treated with IM in association to multimodal analgesia
- ESPB: Erector Spinae Plane Block: Patients treated with ESPB in association to multimodal analgesia

SUMMARY:
This is a prospective observational study conducted at the trauma center of Città della Salute e della Scienza of Turin. The aim of the study is to compare two local regional anesthesia techniques in multimodal analgesia for spine fusion: Intrathecal Morphine (IM) and the Erector Spinae Plane Block (ESPB). The effectiveness of these techniques is to be understood in terms of improved intraoperative and postoperative pain management.

Primary outcome:

● Assessment of postoperative pain upon awakening using the NRS score (T0). The secondary outcomes are aimed at investigating whether one technique is more effective than the other in terms of reducing postoperative opioid consumption and therefore improving pain control in the first 24 hours. Any side effects and complications related to the two techniques will also be analyzed.

Patients are enrolled by signing an informed consent form before surgery. At the time of surgery, an anesthesiologist experienced in locoregional techniques performs one of the two techniques (only those who have been specially trained can perform ESPB). A shared multimodal analgesia protocol is followed intraoperatively. In the postoperative period, standard analgesic therapy is set up and in the first 24 hours parameters, pain (NRS), any rescue medications administered and side effects and complications are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Patients with surgical indication for thoracolumbar spinal fusion with posterior access.
* ASA I, II, III

Exclusion Criteria:

* Patient refusal
* Emergency surgery
* Chronic use (>12 weeks) of opioids in the preoperative period
* Drug addiction
* Contraindication to drugs contained in the protocol
* Contraindications to performing a subarachnoid puncture or fascial block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with presenting surgical indication for thoracolumbar spinal fusion with posterior access. The patients enrolled are being treated at the CTO (Trauma and Orthopedic Center) hospital in Turin.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
NRS score T0 | T0: up to 20 minutes after surgery
  Postoperative pain upon awakening (T0), measured using the NRS (Numeric rating scale) score.

SECONDARY OUTCOMES:
NRS at 2 hours, 4 hours, 6 hours, 12 hours, 24 hours | 2 hours, 4 hours, 6 hours, 12 hours, 24 hours post surgery
  Postoperative pain measured using the NRS score at 2 hours, 4 hours, 6 hours, 12 hours and 24 hours post surgery
Opioid consumption | Consumption of morphine at 2 hours, 4 hours, 6 hours, 12 hours, 24 hours after surgery
  Post-operative opioid consumption (morphine milligram) in the first 24 hours.
Intraoperatory opioid consumption | during the surgery
  Opioid consumption during surgery: intraoperatory remifentanil dosage
Rescue therapy request | During the first 24 hours post surgery
  Time after which the first rescue therapy was requested expressed in hours
Sides effects | First 24 hours after surgery
  Incidence of acute side effects attributable to opioid use (excessive sedation, respiratory depression, nausea and vomiting, pruritus, urinary retention, constipation)
Regional anesthesia complications | Up to first 24 hours after surgery
  Incidence of complications related to subarachnoid puncture or fascial block

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Traumatologico Ortopedico (CTO) - AOU Città della Salute e della Scienza University Hospital, Torino, To, Italy

IPD SHARING:
Plan to Share IPD: Undecided